CLINICAL TRIAL: NCT04531930
Title: Cohort Study on Colorectal Adenoma Canceration in Familial Adenomatous Polyposis
Brief Title: Colorectal Adenoma Canceration in FAP
Status: Not yet recruiting | Type: Observational
Sponsor: Changhai Hospital (Other)
Responsible Party: Principal Investigator, En-Da Yu, Professor, Changhai Hospital
Other Study IDs: SINOFAP2020A
Record Dates: First submitted 2020-08-26; First posted 2020-08-31 (Actual); Last update posted 2020-08-31 (Actual); Status verified 2020-08

CONDITIONS: Familial Adenomatous Polyposis
MeSH Terms: conditions — Adenomatous Polyposis Coli | interventions — Surgical Procedures, Operative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Biospecimen Retention: Samples With DNA — peripheral blood and adenoma samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Surgery Group: Colorectal surgery
  Interventions: Procedure: surgery
- Enhanced Colonoscopy Group: Enhanced colonoscopic treatment and surveillance
  Interventions: Procedure: enhanced colonoscopy
- Self Choice Group: The patients choose the interventional methods, even do nothing.
  Interventions: Other: self choosed methods

INTERVENTIONS:
Procedure: surgery — Colorectal surgery, mainly total proctocolectomy.
  Groups: Surgery Group
Procedure: enhanced colonoscopy — Colonoscopic treatment and surveillance in every 3 months.
  Groups: Enhanced Colonoscopy Group
Other: self choosed methods — A patient chooses a method for himself other than surgery.
  Groups: Self Choice Group

SUMMARY:
The current internationally accepted treatment method for familial adenomatous polyposis is prophylactic total colorectal resection combined with endoscopic follow-up. However, total colorectal resection will bring a sharp decline in the quality of life of patients. Therefore, how to improve treatment methods and improve the quality of life for such patients under the premise of medical quality is the current medical focus. This study intends to establish three parallel observation cohorts, namely the surgical treatment group, the intensive colonoscopy treatment group, and the autonomous monitoring group. During the three-year study period, the investigators observed changes in the number of adenomas, carcinogenesis, and medical expenses in each group during the 3-year study period, and compared the groups to determine whether the intensive colonoscopy therapy has the possibility of delaying or replacing preventive surgery.

DETAILED DESCRIPTION:
Familial adenomatous polyposis is a kind of colorectal cancer syndrome, which belongs to rare diseases. It is estimated that the number of patients in China is about 100,000, accounting for about 1% of all colorectal cancer patients. This type of patients onset between the ages of ten and thirty years old. The typical manifestation is the growth of tens to thousands of colorectal adenomas, and the lifetime risk of colorectal cancer is close to 100%, accompanied by multiple extraintestinal manifestations . Without treatment, the average life span is 40-50 years. The current internationally accepted treatment method is prophylactic total colorectal resection combined with endoscopic follow-up. This program has a significant effect and can extend life expectancy by 10-20 years. However, total colorectal resection will bring a sharp decline in the quality of life of patients. The patients will lose many abilities (working ability, social ability, fertility, etc.) from the age of 20, and the prolonged survival period also brings more misery. This, in turn, also reduces the compliance of treatment. Many patients refuse to accept surgery and turn to endoscopic treatment or even give up treatment. However, there is currently no evidence that methods other than prophylactic surgery can effectively control the risk of colorectal cancer in such patients. Therefore, how to improve treatment methods and improve the quality of life for such patients under the premise of medical quality is the current medical focus. This study intends to establish three parallel observation cohorts, namely the surgical treatment group, the intensive colonoscopy treatment group, and the autonomous monitoring group. Among them, the intensive colonoscopy treatment group will be treated with colonoscopy intensive treatment (that is, colonoscopy treatment is performed every 3 months, Carry out colorectal tumor reduction in segments, and continue to control the growth of adenomas several times) for patients who refuse surgery. During the three-year study period, the investigators observed changes in the number of adenomas, carcinogenesis, and medical expenses in each group during the 3-year study period, and compared the groups to determine whether the intensive colonoscopy therapy has the possibility of delaying or replacing preventive surgery, so as to explore ways to improve the quality of life of such patients.

ELIGIBILITY:
Inclusion Criteria:

* The initial number of polyps is between 100-1000 visually;
* Pathological diagnosis of multiple lesions confirmed colorectal adenoma;
* Germline mutation detection is clearly a point mutation or large deletion of APC gene;
* No cancer or distant metastasis.

Exclusion Criteria:

* Age <18, or >40 years old;
* The initial number of polyps is <100, or >1000;
* The polyp has become cancerous or has suspected distant metastasis;
* Patients with intestinal obstruction, intestinal perforation, intestinal bleeding and other patients who need emergency surgical resection;
* Past history of colorectal surgery;
* Suffering from malignant tumors in other parts and requiring treatment or using chemotherapy drugs or NSAIDs;
* The patient has contraindications to colonoscopy;
* Patients or family members cannot understand the conditions and goals of this study;
* The patient plans to receive surgical treatment of preventive colorectal resection;
* Other reasons considered by the study doctor to be inappropriate for inclusion in the study.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: The anticipants will be allocated in one of the three groups, and accept the corresponding intervention and at least 3 year follow up.
Sampling Method: Probability Sample
Enrollment: 124 (Estimated)
Dates: Start 2020-10-01 (Estimated); Primary Completion 2023-09-30 (Estimated); Study Completion 2030-09-30 (Estimated)

PRIMARY OUTCOMES:
3yCR | 3 years
  3 year Cancerous rate

SECONDARY OUTCOMES:
Adenoma number Change | 3 years
  Change of adenoma number by 3 years
3yOSR | 3 years
  3 year overall survival rate

CONTACTS AND LOCATIONS:
Overall Officials: Jun-Jie XING, MD, Principal Investigator — Changhai Hospital
Locations (1):
- Changhai Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Karstensen JG, Burisch J, Pommergaard HC, Aalling L, Hojen H, Jespersen N, Schmidt PN, Bulow S. Colorectal Cancer in Individuals With Familial Adenomatous Polyposis, Based on Analysis of the Danish Polyposis Registry. Clin Gastroenterol Hepatol. 2019 Oct;17(11):2294-2300.e1. doi: 10.1016/j.cgh.2019.02.008. Epub 2019 Feb 8. PMID 30743005
- [Background] Bulow S. Results of national registration of familial adenomatous polyposis. Gut. 2003 May;52(5):742-6. doi: 10.1136/gut.52.5.742. PMID 12692062